CLINICAL TRIAL: NCT03003260
Title: A Randomized, Double-blind, Cross-over Trial of the Effect of CanChew® Cannabidiol (CBD) Containing Chewing Gum on Patients With Irritable Bowel Syndrome
Brief Title: The Effect of CanChew® Cannabidiol (CBD) Containing Chewing Gum on Irritable Bowel Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Wageningen University (Other)
Responsible Party: Principal Investigator, Renger Witkamp, Head of Nutrition and Pharmacology, Wageningen University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL58588.081.16
Record Dates: First submitted 2016-12-14; First posted 2016-12-26 (Estimated); Last update posted 2016-12-26 (Estimated); Status verified 2016-12

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment A - Treatment B (Experimental): 20 patients receive first 3 weeks treatment A and after a week wash-out 3 weeks treatment B
  Interventions: Other: CBD chewing gum; Other: Placebo
- Treatment B - Treatment A (Experimental): 20 patients receive first 3 weeks treatment B and after a week wash-out 3 weeks treatment A
  Interventions: Other: CBD chewing gum; Other: Placebo

INTERVENTIONS:
Other: CBD chewing gum
  Other Names: CanChew®
Other: Placebo

SUMMARY:
Rationale: IBS is the most common functional gastrointestinal disorder with a prevalence worldwide ranging from 9-23%. Complaints include abdominal discomfort or pain and altered bowel habits. Although the condition is not life-threatening, it strongly impairs quality of life and up to now there is no cure for IBS. It is assumed that IBS symptoms are related to a combination of altered gut motility and secretion, and visceral hypersensitivity. However, its primary cause still remains largely unknown. The endocannabinoid system, together with some functionally related receptors is among the biological targets considered promising for treatment. Modulation of the CB1 , CB2 and related receptors or enzymes of the endocannabinoid system in a broader sense by (endo) cannabinoids or (and) structurally related lipid mediators can influence motility, secretions and decrease hypersensitivity in the gut. Among the plant-derived cannabinoids or so called 'phytocannabinoids', cannabidiol (CBD) is of special interest as it has shown therapeutic potential in preclinical studies and a growing number of case-reports. CBD is a non-specific phytocannabinoid displaying a broad but weak receptor interaction profile. In contrast to the well-known THC from Cannabis sativa, CBD is not psychoactive and often also present in those Cannabis varieties that are not used for their psychoactive properties but for industrial (fibre) or food properties (oil, flour and seeds) instead. Based on preclinical studies and in vitro data we hypothesize that CBD might be able to relieve symptoms of IBS, including pain in patients with IBS. The chewing gum is to be taken 'on demand' and may have some additional perceived positive effects.

Objective: To investigate whether the use of a CBD-containing preparation in the form of CanChew® chewing gum can contribute to a reduction of IBS symptoms and an improvement of perceived wellbeing in patients with IBS.

Study design: A randomized, double-blind, cross-over trial of 8 weeks in total.

Study population: Adults, aged 18-65, diagnosed according to the ROME III criteria with Irritable Bowel Syndrome.

Intervention (if applicable): Patients will, in this cross-over study, receive a maximum 6 chewing gums per day, either containing 50 mg of cannabidiol per chewing gum in case of the CanChew chewing gum, or a placebo chewing gum. This first intervention period will last 3 weeks. Next, participants will undergo a one week wash-out and then switch intervention to either placebo or the CanChew chewing gum for another 3 weeks.

Main study parameters/endpoints: The main study parameter is a change in pain reduction perception experienced and measured by the patient using VAS-scales before and after taking the chewing gum, to be recorded in a diary. Next to this a patient is asked to provide one VAS score for each completed week. Furthermore, the adequate relief will be measured every day. At the end of each week patients will also be asked (from their diary) whether they noticed a change in stool frequency or (and) experienced any side-effects. For the disease-related quality of life the IBS-QOL will be used. This questionnaire will be filled out in week 1, 4, 5, and 8.

ELIGIBILITY:
Inclusion Criteria:

* Male
* Female, only when using the contraceptive pill
* Adults, aged 18-65
* IBS, diagnosed according to the Rome III criteria
* More than 3 moments of pain with a vas-score of 4 and higher per week
* Signed informed consent

Exclusion Criteria:

* Use SSRIs, tramadol or tramagetic
* Have a history of intestinal surgery that might interfere with the outcome of the study
* Female patients: currently pregnant or breast-feeding hope to become pregnant during the study, judged by the persons self.
* Female who is not using the contraceptive pill.
* Are an employee and students of the department of Human Nutrition at Wageningen UR, or employee at the MDL department of hospital Gelderse Vallei
* Participate in another research study
* Alcohol use (male more than 14 servings a week, female more than 7 servings a week)
* Cannabis use is from 3 months before until the end of the study not allowed.
* Hypersensitivity to one of the ingredients of the chewing gum
* Drug use (CYP2C19 and CYP3A4) metabolised; medication will be evaluated for this by the principal and medical investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-12; Primary Completion 2017-04 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Change of pain scores on the Visual analoge scale (VAS) between baseline and 3, 5 and 8 weeks of treatment | Baseline, 3 weeks, 5 weeks and 8 weeks
  The main study parameter is a change in pain reduction perception experienced and measured by the patient using VAS-scales before and after taking the chewing gum, to be recorded in a diary

SECONDARY OUTCOMES:
Change of IBS-QOL baseline vs 3, 5 and 8 weeks of treatment | Baseline, 3 weeks, 5 weeks and 8 weeks
  For the disease-related quality of life the IBS-QOL will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No